CLINICAL TRIAL: NCT03684252
Title: Reducing Self-stigma in Persons With HIV and Drug Use Disorders in Primary Health Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Responsible Party: Principal Investigator, Coralee Perez-Pedrogo, Principal Investigator, University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A3890118
Record Dates: First submitted 2018-09-14; First posted 2018-09-25 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Drug Use Disorders; HIV/AIDS
Keywords: Self-stigma; Drug Use Disorders; HIV
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Treatment as usual
  Interventions: Other: Treatment as Usual
- Intervention (Experimental): CBT-based intervention
  Interventions: Behavioral: CBT-based intervention

INTERVENTIONS:
Behavioral: CBT-based intervention — Cognitive Behavioral Therapy (CBT) that uses acceptance and mindfulness strategies, together with commitment and behavior change strategies.
  Arms: Intervention
Other: Treatment as Usual — Participants' will receive treatment as usual.
  Arms: Control

SUMMARY:
The investigators propose to lay the groundwork for a larger effectiveness clinical trial that will lead to the advancement of a novel evidence-based treatment for DUD and HIV among Spanish-speaking Latinos who suffer from self-stigma and have inadequate treatment adherence. This pilot project aims to: compare the outcomes of a culturally adapted CBT-based intervention to treatment as usual (TAU), in a randomized pilot trial of HIV+ individuals with a lifetime DUD.

DETAILED DESCRIPTION:
This treatment model, new for Puerto Rico, should improve compliance with ART and health outcomes for Latino patients who have largely been excluded from efficacy and effectiveness studies, and thus have not benefited from these advances. The proposed research lays the groundwork to provide the benefits of theoretically grounded, culturally adapted, and evidence-based treatment to reduce self-stigma and increase drug and HIV treatment adherence among Puerto Ricans that may also apply to other Spanish-speaking patients.

The investigators work is guided by the Stage Model for Behavior Therapy that recognizes that the scientific study of behavior therapies involves a systematic developmental process that progresses from feasibility (Stage I) to efficacy (Stage II) to effectiveness (Stage III). The proposed research focuses on Stage Ib where the investigators propose to conduct a pilot randomized control trial to compare the outcomes between a novel CBT-based intervention and treatment as usual (TAU) among HIV/DUD+ Latinos reporting self-stigma who are receiving care in a primary care health setting. Assessments of self-stigma and HIV and drug treatment adherence for all participants will be collected pre-treatment and post-treatment. This model allows to lay the groundwork for a larger effectiveness clinical trial.

The investigators plan to enroll 16 patients who will be randomly assigned to the CBT (n=8) or to TAU (n=8). Sample size considers a 35% attrition rate as based in previous research experiences among similar population. Patients will be recruited in primary health care clinics in PR. Participants will be randomly assigned to (a) treatment as usual or (b) a Cognitive and Behavioral Therapy. This intervention is a theoretically-based efficacious treatment for self-stigma and related depression. It consists of weekly 60-minute sessions for 6-8 weeks; is flexible and can be modified to fit the needs of individual clients. The intervention is designed to help individuals to employ acceptance and values-directed behavior change strategies in order to increase psychological flexibility, a process that is at the core of behavioral health and retention in treatment.

Overall, analyses will allow generating an effect size that can be used to calculate the number of subjects needed for adequate power to detect significant differences between groups.

ELIGIBILITY:
Inclusion Criteria:

Spanish speakers that comply with

* A drug use disorder based on the Spanish version of the short form of the WHO Composite International Diagnostic Interview (CIDI) that has been used widely in Puerto Rico;
* HIV clinical criteria;
* Moderate to higher levels of HIV felt self-stigma (>25);
* Using the clinic as the main source of medical care during the study; and
* Agreement to random assignment

Exclusion Criteria:

* DUD/HIV+ individuals who are not prescribed ART;
* An acute medical emergency (physical or psychiatric),
* Unable to provide informed consent
* Who are actively suicidal.
* Cognitive impairment or dementia based on a score of 24 or less on the Mini Mental State Examination

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Substance Abuse Self-stigma Scale (change is being assessed) | Change from baseline/pre-treatment at any point from last intervention (for both groups) to up to 2 weeks after
  Psychometrically sound and culturally adapted, this is a 40-item scale that contains four sub-scales that measures self-devaluation, fear of enacted stigma, stigma avoidance, and values disengagement due to self stigma. Internal consistency coefficients for the sub-scales ranged from .82 to .88. Study participants will need to endorse at least three items from the self-devaluation sub-scale to be considered as presenting self-stigma (this will be used as an inclusion criteria). Item endorsement will be analyzed as a count, per sub-scale. The greater number of items endorsed per sub-scale, will be indicative of a higher level of self-stigma as manifested by the sub-scale construct.

SECONDARY OUTCOMES:
HIV Felt-stigma Scale (change is being assessed) | Change from baseline/pre-treatment at any point from last intervention (for both groups) to up to 2 weeks after
  The scale measures felt and enacted stigma constructs among persons living with HIV (PLWHIV). Developed for Spanish-speaking populations, this is a 17-item, self-administered multi-dimensional measure for felt and enacted stigma in PLWHIV, using a 4-point Likert scale and that is culturally-sensitive. Exhibits adequate alpha and Pearson correlation coefficients (0.91 and 0.68, respectively) and convergent validity. The scale has four dimensions which scores will be summed to obtain a total scale score. The total scale score is indicative of the level of HIV-related felt stigma experienced by a person. Scale ranges are interpreted as follows: 0-15 no stigma; 16-24 mild; 25-35 moderate; and > 35 severe. For this study, a total score of > 25 is required for enrollment.
Depressive symptoms (change is being assessed) | Change from baseline/pre-treatment at any point from last intervention (for both groups) to up to 2 weeks after
  To assess depressive symptoms, the study will use The Patient Health Questionnaire, depression module: Is a 8 item validated measure. The Spanish version showed a sensitivity of 77% and a specificity of 100% when compared to the Structured Clinical Interview for DSM mood module. The higher the score obtained on the scale, the greater the manifestation of depressive symptoms.
Adherence to Combination Therapy Questionnaire (change is being assessed) | Change from baseline/pre-treatment at any point from last intervention (for both groups) to up to 2 weeks after
  The research team have completed translation, back-translation, and agreements with an expert/bilingual panel of the Single-Item Self-Rating Adherence Scale (SRSI). This is a single item scale that has been use successfully among the health sector.

CONTACTS AND LOCATIONS:
Overall Officials: Coralee Perez-Pedrogo, PhD, Principal Investigator — University of Puerto Rico
Locations (1):
- University of Puerto Rico Medical Sciences Campus, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No